CLINICAL TRIAL: NCT05993520
Title: Effects of Respiratory Muscle Functions on Interstitial Lung Disease: Sleep Quality, Dyspnea, and Fatigue
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Collaborators: TURK TORAKS DERNEGI (Unknown)
Responsible Party: Principal Investigator, Goksen Kuran Aslan, Associate professor, Istanbul University - Cerrahpasa
Other Study IDs: GAslan-2023
Record Dates: First submitted 2023-07-21; First posted 2023-08-15 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Interstitial Lung Disease
Keywords: Interstitial Lung Disease; Respiratory Muscles; Sleep; Quality of Life; Fatigue
MeSH Terms: conditions — Lung Diseases, Interstitial; Fatigue | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interstitial Lung Disease: Between June 2020 and June 2023, a total of 36 voluntary participants, aged 18 and above, who were receiving treatment at the Department of Chest Diseases, Istanbul Faculty of Medicine, Istanbul University, and met the inclusion criteria, were included in the study.
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Between June 2020 and June 2023, 36 volunteer participants aged 18 and above, who were receiving treatment in the Department of Chest Diseases at Istanbul University, Istanbul Faculty of Medicine, and met the inclusion criteria, were included in the project. Participants' respiratory function tests, respiratory muscle functions, dyspnea levels, cough, sleep quality, peripheral muscle strength, quality of life, exercise capacity, and fatigue levels were evaluated.

SUMMARY:
Although there are numerous data demonstrating the impact of Interstitial Lung Disease (ILD) on respiratory functions, there is a lack of studies investigating the effects of respiratory functions on parameters such as sleep quality, dyspnea, and fatigue. The primary objective of the study is to examine the influence of changes in respiratory muscle functions in ILD on sleep quality, dyspnea, and fatigue parameters. The secondary objective is to investigate the effects of respiratory muscle functions in ILD on parameters such as cough, pain, exercise capacity, peripheral muscle strength, anxiety, depression, and quality of life.

DETAILED DESCRIPTION:
Introduction: Despite having numerous data demonstrating the impact of Interstitial Airway Disease (IAD) on respiratory functions, there is a lack of studies investigating the effects of respiratory functions on parameters such as sleep quality, dyspnea, and fatigue. The primary objective of the study is to examine the effects of changes in respiratory muscle functions in IAD on sleep quality, dyspnea, and fatigue parameters. The secondary objective is to investigate the effects of respiratory muscle functions in IAD on parameters such as cough, pain, exercise capacity, peripheral muscle strength, anxiety, depression, and quality of life.

Methods: Between June 2020 and June 2023, 36 volunteer participants aged 18 and above, who were receiving treatment in the Department of Chest Diseases at Istanbul University, Istanbul Faculty of Medicine, and met the inclusion criteria, were included in the project. Participants' respiratory function tests, respiratory muscle functions, dyspnea levels, cough, sleep quality, peripheral muscle strength, quality of life, exercise capacity, and fatigue levels were evaluated. Pearson Correlation Test was applied to determine the relationship between variables. Multiple linear regression analysis was used to examine factors that could affect respiratory muscle strength and endurance values.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older.
* Having a diagnosis of Interstitial Lung Disease (ILD) by a chest diseases specialist.

Exclusion Criteria:

* Systemic involvement of ILD
* Cooperation problem
* Presence of orthopedic/neurological issues hindering walking and exercise.
* Uncontrolled cardiovascular disease.
* Presence of acute upper and lower respiratory tract infections.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Between June 2020 and June 2023, a total of 36 voluntary participants, aged 18 and above, who were receiving treatment at the Department of Chest Diseases, Istanbul Faculty of Medicine, Istanbul University, and met the inclusion criteria were included in the study.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
sleep quality-1 | 5 minutes
  Pittsburgh Sleep Quality Index (PSQI) will be used to assess sleep quality. PSQI is a scale consisting of 24 questions that evaluate sleep quality and disturbances in the past month. Each item is scored between 0 and 3, and a total score higher than 5 indicates insufficient sleep quality in the individual.
Sleep Apnea | 5 minutes
  Obstructive Sleep Apnea Syndrome Risk: The STOP-BANG questionnaire will be used to assess the risk of Obstructive Sleep Apnea Syndrome (OSAS). The questionnaire consists of a total of eight questions that are answered with "yes" or "no." In the STOP section of the questionnaire, if at least two out of the four questions are answered "yes," it is considered a high risk for OSAS.
Modified Medical Research Council Questionnaire | 5 minutes
  To assess dyspnea, the Modified Medical Research Council (mMRC) Questionnaire will be used.
  The mMRC is a scale used to assess the level of dyspnea during daily life activities. It involves a five-point category scale (0 to 4) in which patients choose the expression that best describes their level of dyspnea. As the score increases, the severity of dyspnea also increases.
Dyspnea-12 Scale | 5 minutes
  To assess dyspnea, the Dyspnea-12 Scale will be used.
  The Dyspnea-12 Scale is a 12-item questionnaire that measures the intensity of dyspnea. It consists of a four-point Likert-type scale (0=none, 1=mild, 2=moderate, 3=severe) as response options.The minimum score is 0, and the maximum score is 36. An increase in the score indicates an increase in the severity of dyspnea experienced by the patient.
fatigue | 5 minutes
  For the assessment of fatigue, the Fatigue Assessment Scale (FAS) will be used. The FAS is a subjective fatigue questionnaire consisting of 10 items. It utilizes a five-point Likert scale (1=Always-5=Never) as response options. The total scores that can be obtained from the FAS range from 10 to 50. Higher scores indicate a higher level of fatigue experienced by the individual.
Respiratory Function Test | 5 minutes
  Respiratory Function Test: The respiratory function status of patients will be assessed using spirometric testing.Spirometry is a medical test used to assess the functioning of the lungs. It measures the amount of air a person can inhale and exhale, as well as the speed and volume of airflow. This test is essential for diagnosing and monitoring lung conditions such as interstitial lung disease, chronic obstructive pulmonary disease (COPD), and other respiratory disorders.The spirometry results are compared to predicted values based on factors such as age, height, sex, and ethnicity. This comparison helps healthcare professionals identify any deviations from normal lung function.
Respiratory Muscle Strength | 5 minutes
  Respiratory Muscle Strength: The easiest and most common method is measuring mouth pressure during voluntary contraction against a closed airway to open the airway. In the study, respiratory muscle strength will be evaluated using the "Vyaire Medical MicroRPM" device. Maximum Inspiratory Pressure (MIP): At least three measurements are taken, and the highest value is recorded. Maximum Expiratory Pressure (MEP): The best of at least three measurements is recorded.
Comorbidity | 3 minutes
  Charlson Comorbidity Index: It is a widely used index in clinical practice that queries chronic systemic diseases, assesses their frequency and relationships. It consists of nineteen different items. The scores obtained from the patient's comorbid conditions are added together to obtain a score, and a score is also added based on the patient's age. This age score is 1 for ages 50-59, 2 for ages 60-69, 3 for ages 70-79, 4 for ages 80-89, and 5 for ages 90-99.
Respiratory Muscle Endurance: | 8 minutes
  Respiratory Muscle Endurance: In respiratory muscle endurance measurement, an incremental threshold load test will be applied using the "Threshold IMT" device. According to the incremental threshold load protocol, after determining the MIP value, the threshold pressure is set at approximately 20-40% of MIP. The threshold pressure is increased every two minutes. The highest pressure that the patient can sustain for at least one minute is recorded as the patient's respiratory muscle endurance value.

SECONDARY OUTCOMES:
Cough | 5 minutes
  Leicester Cough Questionnaire will be used for the assessment of cough. It consists of 19 items with a 7 point likert response scale (range from 1 to 7).Each item is developed to assess symptoms during cough and impact of cough on three main domains: physical, psychological and social. Scores are calculated as a mean of each domain and the total score is calculated by adding every domain score. The total severity score ranges 3-21, with a lower score indicating greater impairment of health status due to cough.
Symptoms Seveerity | 1 minutes
  Dispnea, Pain, and Cough Severity: Dispnea, pain, and cough severity will be assessed using the Visual Analog Scale (VAS). VAS is used to convert some values that cannot be measured numerically into numerical form. It involves a 100 mm line with the two endpoints representing the two extreme definitions of the parameter to be evaluated (e.g., no pain/cough - very severe pain/cough). The patient is asked to indicate their own condition by drawing a line, placing a dot, or marking a point on this line to indicate where their situation corresponds. The point marked by the patient is measured using a ruler. The resulting number represents the patient's level of pain/cough severity.
exercise capacity | 8 minutes
  The Six-Minute Walk Test (6MWT) will be used to assess exercise capacity. The 6MWT determines individuals' submaximal functional exercise capacity. The patient will be asked to walk as far as possible at their own walking pace for six minutes in a straight 30-meter corridor. Before starting the test, the patient rests in a sitting position in the corridor for 10 minutes. Prior to the test, oxygen saturation, heart rate, blood pressure, dyspnea, and leg fatigue scores are recorded using the Modified Borg Scale. If the patient wants to rest during the test, the resting time is included in the test duration without stopping the stopwatch. At the end of the test, the assessments made before the test are repeated. The distance walked in six minutes (6MWD) is recorded in meters.
peripheral muscle strength | 5 minutes
  The "J-Tech CommanderTM Muscle Tester" hand-held dynamometer will be used to assess the strength of the quadriceps femoris muscle. The hand-held dynamometer is a simple, easy-to-use, portable, time-efficient, inexpensive, and lightweight device that measures maximum isometric muscle strength.
anxiety&depression | 5 minutes
  The Hospital Anxiety and Depression Scale (HADS) will be used to determine the anxiety and depression status. HADS is a self-report questionnaire developed to assess the risk, level, and severity of anxiety and depression in individuals with physical illnesses and those seeking primary healthcare services. It consists of a total of 14 questions, with seven questions (odd numbers) measuring anxiety and the other seven questions (even numbers) measuring depression. It is a four-point Likert-type scale. The cutoff score for the anxiety subscale (HADS-A) is 10/11, and for the depression subscale (HADS-D) is 7/8.
health problems | 5 minutes
  The Nottingham Health Profile (NHP) was originally created as a standardised tool to survey health problems and measure medical or social interventions. The NHP is a patient-reported questionnaire. Respondents tick yes or no boxes to answer questions about their health and its effects on their daily life.
  The questionnaire is divided into two parts. The first parts comprises 38 questions in six categories: sleep, physical mobility, energy, pain, emotional reactions, and social isolation. This first section is weighted to reflect how severe an impact the respondent thinks their health is having on the above areas of life. The second part of the NHP is made up of seven statements about areas of life that are commonly affected by health: paid employment, jobs around the house, social life, personal relationships, sex life, hobbies and interests, and holidays. Scores on the NHP can range from 0 i.e. no distress to 100 i.e severe distress.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Üniversitesi-Cerrahpaşa, Istanbul, Buyucekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bloem AEM, Houben-Wilke S, Mostard RLM, Stoot N, Janssen DJA, Franssen FME, Custers JWH, Spruit MA. Respiratory and non-respiratory symptoms in patients with IPF or sarcoidosis and controls. Heart Lung. 2023 Sep-Oct;61:136-146. doi: 10.1016/j.hrtlng.2023.05.013. Epub 2023 Jun 2. PMID 37269615